CLINICAL TRIAL: NCT05925673
Title: Early Neuromuscular Stimulation and Mirror Therapy Interventions During Immobilization of Distal Radius Fracture
Brief Title: Early NMES and Mirror Therapy Interventions During Immobilization of Distal Radius Fracture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Western University (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Joy MacDermid, Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 120275
Record Dates: First submitted 2023-06-20; First posted 2023-06-29 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Distal Radius Fracture
Keywords: Neuromuscular Stimulation; Mirror Therapy; Early Intervention
MeSH Terms: conditions — Wrist Fractures | interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard of Care (No Intervention): Participants will follow standard practice protocols at the Roth McFarlane Hand and Upper Limb Centre in London.
- Mirror Therapy (Experimental): Participants will engage in a home based mirror therapy intervention from 3 to 6 weeks post-fracture.
  Interventions: Other: Mirror Therapy
- Neuromuscular Stimulation (NMES) (Experimental): Participants will engage in a home based neuromuscular stimulation intervention from 3 to 6 weeks post-fracture.
  Interventions: Other: Neuromuscular Stimulation (NMES)
- Mirror Therapy + NMES (Experimental): Participants will engage in a home based combined mirror therapy + neuromuscular stimulation intervention from 3 to 6 weeks post-fracture.
  Interventions: Other: Mirror Therapy + NMES

INTERVENTIONS:
Other: Mirror Therapy — Participants will perform exercises with their unaffected arm in front of a mirror with the affected arm hiding behind the mirror. They will watch the reflection of the unaffected arm as they perform the exercises to provide visual feedback that the affected arm is performing the exercises. They will repeat this procedure for 10 minutes, 3 times a day, 5 days a week for 3 weeks.
  Arms: Mirror Therapy
Other: Neuromuscular Stimulation (NMES) — Participants will use a portable NMES machine to stimulate the wrist extensors and flexors of the affected arm at a low intensity with the arm relaxed. They will repeat this procedure for 10 minutes, 3 times a day, 5 days a week for 3 weeks.
  Arms: Neuromuscular Stimulation (NMES)
Other: Mirror Therapy + NMES — Participants will perform exercises with their unaffected arm in front of a mirror with the affected arm hiding behind the mirror. They will watch the reflection of the unaffected arm as they perform the exercises to provide visual feedback that the affected arm is performing the exercises. During the exercises they will have a portable NMES machine set up to stimulate the wrist extensors and flexors of the affected arm at a low intensity with the arm relaxed. They will repeat this procedure for 10 minutes, 3 times a day, 5 days a week for 3 weeks.
  Arms: Mirror Therapy + NMES

SUMMARY:
Current practice for distal radius fractures is to begin rehabilitation after immobilization to remediate the resulting impairments. Neuromuscular electrical stimulation and mirror therapy are strategies that integrate neurological and musculoskeletal activation, that may be beneficial for mitigating the resulting impairments if applied during immobilization. The study aim is to determine whether neuromuscular stimulation and mirror therapy interventions can be implemented during immobilization for distal radius fractures to minimize the resulting impairments when compared to standard rehabilitation.

DETAILED DESCRIPTION:
Distal radius fractures are one of the most common orthopedic injuries require 6 to 8 weeks of immobilization for bone healing making it an ideal model to evaluate the negative consequences of immobilization. Consequences of immobilization include motor dysfunction (e.g. muscular atrophy), loss of the representation of motor and sensory function, and loss of fine motor skills. Current practice is to begin rehabilitation after immobilization to remediate these impairments. Neuromuscular electrical stimulation and mirror therapy are strategies that integrate neurological and musculoskeletal functioning, that can be used during immobilization to mitigate negative consequences. To date, these strategies have primarily been implemented in stroke rehabilitation, but minimal research has been done to assess their effectiveness with musculoskeletal populations. The study aim is to determine whether neuromuscular stimulation and mirror therapy interventions can be implemented during immobilization for distal radius fractures to minimize impairments when compared to standard rehabilitation. Four groups will be compared: group 1 will engage in standard care, group 2 will engage in a mirror therapy intervention during immobilization, group 3 will engage in a neuromuscular stimulation intervention during immobilization, and group 4 will engage in a combined mirror therapy + neuromuscular stimulation intervention during immobilization. Patient reported and objective outcome measures will be assessed at baseline (before starting intervention; 3 weeks), after cast removal and completion of the intervention (6 weeks), 8 (to 10) weeks, and 12 weeks post fracture. Ideally these interventions will improve outcomes and facilitate rehabilitation after distal radius fracture which could allow patients to return to their daily activities and work more readily after fracture.

ELIGIBILITY:
Inclusion Criteria:

* Sustained a distal radius fracture in the last 3 weeks being managed conservatively in a cast
* Able to understand instructions in English
* Able to give informed consent (no known cognitive impairment that would limit this)

Exclusion Criteria:

* Cognitive disorders that would preclude the participant from following instructions and engaging in the home interventions
* Visual impairments that limit ability to engage in NMES and mirror therapy interventions
* Superficial metal implants in the injured arm
* Cancer (active)
* Severe peripheral vascular disease
* Thrombophlebitis in injured arm

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-02-09 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Adherence | 6 weeks post fracture
  % of sessions completed

SECONDARY OUTCOMES:
Patient-Rated Wrist Evaluation (PRWE) | Baseline, 6, 8 to 10, and 12 weeks post fracture
  Participants will report their pain for 5 items, their function for 10 items on a scale from 0 (Never) to 10 (Always). The overall score (sum of pain + function sub scales) is out of 150, with a higher score representing more pain and disability.
EuroQol-5D (EQ-5D) | Baseline, 6, 8 to 10, and 12 weeks post fracture
  Participant rates their health status from 0 (the worst health you can imagine) to 100 (the best health you can imagine). The higher the score, the better the health status.
Single Assessment Numeric Evaluation (SANE) | Baseline, 6, 8 to 10, and 12 weeks post fracture
  On a scale from 0 to 100. with 100 being normal, participants rate the function of their wrist on that day. A higher score represents better function.
Global Rating of Change (GRC) | Baseline, 6, 8 to 10, and 12 weeks post fracture
  Participants will rate the overall condition of their elbow/wrist from when they started treatment until the point of measurement on a scale of -5 (very much) to 5 (completely recovered). The higher the score the greater the improvement.
Numeric Pain Rating Scale (NPRS) at rest | Baseline, 6, 8 to 10, and 12 weeks post fracture
  Participants will rate their pain level at rest on a scale from 0 (no pain) to 10 (unbearable pain).
Range of motion (ROM) - unaffected side | Baseline, 6, 8 to 10, and 12 weeks post fracture
  Wrist flexion, extension, ulnar deviation, radial deviation, elbow supination, elbow pronation, and thumb extension (radial abduction of the thumb) will be measured using a goniometer with the participant in a seated position and their arm by their side. Wrist movements will be measured with the elbow at a 90 degree angle. ROM will be recorded as degrees of motion. Higher scores will represent greater ROM.
Range of motion (ROM) - affected side | 6, 8 to 10, and 12 weeks post fracture
  Wrist flexion, extension, ulnar deviation, radial deviation, elbow supination, elbow pronation, and thumb extension (radial abduction of the thumb) will be measured using a goniometer with the participant in a seated position and their arm by their side. Wrist movements will be measured with the elbow at a 90 degree angle. ROM will be recorded as degrees of motion. Higher scores will represent greater ROM.
Dexterity | Baseline, 6, 8, 10, and 12 weeks post fracture
  Dexterity will be measured using a Purdue Pegboard. Participants will be seated at a table with the Purdue Pegboard in front of them. They will complete four subtests. First they will place as many pins as they can in the holes with the right hand in 30 sec. This will be repeated on the left. For the third condition they will have 30 sec to place as many pins in the holes using both hands simultaneously. The final condition they will assemble the pins, washers, collars, and washers leading with one hand for 60 sec, then repeating with the other hand leading for 60 sec. For each condition they will be instructed to complete as many as possible in the allotted time. Higher scores indicate better dexterity. During baseline assessment only the single hand condition for the unaffected side will be assessed.
Vividness of Movement Imagery Questionnaire-2 (VIMQ-2) | Baseline, 8 to 10, and 12 weeks post fracture
  A 36-item questionnaire with twelve actions that are imagined kinaesthetically and from an internal and external visual perspective. The vividness of each imagination is rated on a scale from 1 (Perfectly clear and as vivid (as normal vision or feel of movement)) to 5 (No image at all, you only "know" that you are thinking of the skill). Scores range from 36 to 180, with lower scores indicative of vivid imagery.
Pinch Strength - unaffected side | Baseline, 6, 8 to 10, and 12 weeks post fracture
  Pinch grip will be measured in pounds using a Jamar Hydraulic Pinch Gauge with the participant in a seated position with their elbow resting on a table. Higher scores will represent a stronger pinch grip.
Pinch Strength - affected side | 8 to 10, and 12 weeks post fracture
  Pinch grip will be measured in pounds using a Jamar Hydraulic Pinch Gauge with the participant in a seated position with their elbow resting on a table. Higher scores will represent stronger pinch grip.
Electromyography (EMG) | 8 to 10 and 12 weeks post fracture
  Electromyography of the wrist flexors and extensors will be measured using the DELSYS Trigno Wireless Biofeedback System. EMG will be assessed during the three maximum voluntary contractions (MVC) for 5 sec in wrist flexion, radial deviation, wrist extension, and ulnar deviation on both sides. Participants will be seated with their arm by their side and elbow at a 90 degree angle. For wrist flexion and radial deviation, participants will have their hands under the table to push up into it for the MVC. With wrist flexion the palm is facing the ceiling and for radial deviation their hand will make a fist with their thumb oriented towards the ceiling. For wrist extension and ulnar deviation, participants will have their hand set on top of the table to push down into it for the MVC. For wrist extension, their fingers will be extended and palm facing the ceiling. For ulnar deviation, participants will make a fist and their thumb will be oriented towards the ceiling.
Grip Strength - unaffected side | Baseline, 6, 8 to 10, and 12 weeks post fracture
  Grip strength will be measured with the patient in a seated position with their elbow resting on a table. A Jamar Hydraulic Hand Dynamometer will be used as a means to measure grip strength in pounds. Higher scores will represent greater grip strength.
Grip Strength - affected side | 8 to 10, and 12 weeks post fracture
  Grip strength will be measured with the patient in a seated position with their elbow resting on a table. A Jamar Hydraulic Hand Dynamometer will be used as a means to measure grip strength in pounds. Higher scores will represent greater grip strength.
Numeric Pain Rating Scale (NPRS) during movement | Baseline, 6, 8 to 10, and 12 weeks post fracture
  Participants will rate their pain level during movement on a scale from 0 (no pain) to 10 (unbearable pain).

CONTACTS AND LOCATIONS:
Overall Officials: Joy MacDermid, PhD, Principal Investigator — Western University
Locations (1):
- Roth | McFarlane Hand and Upper Limb Center, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No